

# <u>APPENDIX 1 – PATCHS SCREENSHOTS (INCLUDING PARTICIPANT CONSENT</u> FORM)

## IMPROVING THE ACCURACY OF ARTIFICIAL INTELLIGENCE TRIAGE IN PRIMARY CARE

### (AI TRIAGE ACCURACY)

### **Version history**

| 1 | | |
|---|---|---|
| Version | Date | Summary of changes |
| 1.0 | 2023-08-10 | Initial draft |
| 1.1 | 2025-05-16 | Screenshot 9 updated to reflect the current Patchs design |
| 1.2 | 2025-09-03 | Screenshots 9 and 10 updated to include a link to further information on |
| | | approved research studies. Screenshot 11 added. |



Screenshot 1: Triage decisions made by GP practice staff



Screenshot 2: Triage decisions pre-populated by Patchs AI



### Hide ^ Triage decision How clinically urgent is this message? Help ✓ O Routine Urgent O Emergency O Admin / Med request This urgency was chosen by PATCHS AI . Change it if you disagree. What are the main topics of this message? (Optional) Help 🗹 Add another topic... Back Pain 😮 This topic was chosen by PATCHS AI . Change it if you disagree. *Ideally*, who do you think *should have* dealt with this message? Help 🗹 Choose... What actions are required from you to resolve this message? Help Z ☐ Give patient information (e.g. advice) ☐ Fill out paperwork (e.g. Med 3, TWIMC letter) Order tests (e.g. blood tests, X-ray) Telephone patient Prescribe new medication Video call patient Re-authorise / issue repeat medication See patient face-to-face ☐ Visit patient at home Signpost to another service (e.g. IAPT, physio) Mark as duplicate (e.g. if patient chasing) This action was chosen by PATCHS AI . Change it if you disagree.

### Screenshot 3: Urgency AI - prioritises online consultations in inbox



Screenshot 4: Topic AI – example asking further questions





### Screenshot 5: Assign AI – assigns online consultations to a 'Clinical' inbox







Screenshot 7: Signpost AI – example emergency message



Based on the information you have entered, you may need emergency medical help. If this is a <u>medical emergency</u> you should cancel this request and call 999, or go to your <u>local A&E</u> immediately.

Click the links below for information from the NHS related to your query. (Please note, some may not be relevant.)

• Stroke

Would you still like to submit your request to your GP practice at your own risk?

Please be aware that if you submit your request to your GP practice, your request may not be dealt with quickly enough, or with the right treatment you need, which could result in your injury or death. 'At your own risk' means that if this happens you accept it will be your responsibility, and not the responsibility of your GP practice.

1 message remaining.

No, I will call 999 or go to A&E

Yes, I would still like to contact my GP practice at my own risk

#### Screenshot 8: Signpost AI – example routine message

Click the links below for information from the NHS related to your query. (Please note, some may not be relevant.)

• Hair Loss

Would you still like to submit your request to your GP practice?

1 message remaining.

No, this information has resolved my query

Yes, I would still like to contact my GP practice



# Screenshot 9: Notice when patients or their carers use PATCHS that their anonymised data may be shared with The University of Manchester for research purposes



Health Hub

Patchs GP

Help



### **Langworthy Medical Practice**

### Create an account to contact your GP online

Patchs is a service provided by your GP practice to help them care for their patients. Read more about Patchs 🗹

Patchs Health is the trading name of Spectra Analytics Limited company number 09108913. Patchs Health processes your data under their Legitimate Interest for quality and assurance purposes, for the benefit of patients and GP practices.

We anonymise data we collect. 'Anonymised' means you cannot be identified. Information such as name, address, and date of birth are removed. Anonymised data may include information such as your age, sex, ethnicity, and medical information. This may be shared with researchers (such as the University of Manchester) and external GPs evaluating the software's safety and effectiveness. Anonymised data will be retained for 5 years after it has finished being used. At any time, you can stop sharing your anonymised data with researchers on the 'Data Privacy' page in the top menu after creating an account and logging in.

To see a list of NHS-approved research studies using anonymised Patchs data please visit this page 🗹.

For further information on how we process data and our compliance with data protection law please visit our privacy policy 🗹.

It is important that you read and understand the terms and conditions in the End User License Agreement 🗹 before continuing. By pressing the 'Accept and continue' button below you confirm you are 16 years or older and have read, understood, and accept the terms and conditions in the End User License Agreement 🗹 .

Accept and continue





#### Screenshot 10: Opt-out toggle button in PATCHS that patients can access at any time





### Screenshot 11: Page showing list of NHS-approved research studies using anonymised Patchs data

PATCHS Support / GP practices / General information on Patchs / Research evidence

# NHS-approved research studies using anonymised Patchs data



### **Al Triage Accuracy**

Full title: Improving the accuracy of artificial intelligence triage in primary care

**IRAS ID: 331286** 

**Chief Investigator:** Dr Benjamin C Brown (University of Manchester). Dr Brown is a part-time employee of Patchs Health as Chief Medical Officer and is a shareholder in the company. Patchs Health develop the Patchs software.

Contact email: patchs.research@manchester.ac.uk

Sponsor organisation: University of Manchester

#### Research summary:

WHY ARE WE DOING THIS?

When patients contact their GP practice, the first step is to work out what kind of help they need and how quickly it's needed. This is called 'triage' and is important for patient safety. Artificial Intelligence (AI) can help make triage faster. While AI is already being used in the NHS, we don't know how accurate it is or if it treats all patients fairly.

WHAT WILL WE DO?

We will collect anonymised data from patients that use an AI triage system called Patchs in GP practices in England. The project will last four years. We will analyse the data in four steps:

- 1. Look at data from GP practices using Patchs without AI triage to see how they currently triage patients and what problems they face.
- 2. Use data from GP practices using Patchs (both with AI on and off) to make the AI triage more accurate.
- 3. Check data from GP practices using Patchs with AI triage off to measure how well the updated AI system works.



- 3. Check data from GP practices using Patchs with AI triage off to measure how well the updated AI system works.
- 4. Give the improved AI triage system to GP practices already using AI.

At each step, we will check whether patients from different backgrounds are treated fairly.

HOW WILL WE ANALYSE THE DATA?

We will use statistical methods to compare the triage decisions made by the AI with those made by clinical staff. This analysis will also be used to check that the AI works fairly for patients from different backgrounds.

WHAT DIFFERENCE WILL WE MAKE?

Our research will show the problems with triage and explain how an improved AI system could help patients get the care they need more quickly.

Research Ethics Committee name: Nottingham 1 REC

REC reference: 25/EM/0191

Date of REC Opinion: 01 Aug 2025

Was this article helpful?

Yes No